CLINICAL TRIAL: NCT03561077
Title: Feasibility in France of a Mindfulness-based Group Therapy for Adolescents With Chronic Pain
Acronym: PEACEFULL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0354; 2017-A03338-45 (Other: ID-RCB)
Record Dates: First submitted 2018-04-27; First posted 2018-06-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain
Keywords: Pain; Pediatrics; Mindfulness; Adolescents
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness program (Experimental): To study the feasibility in France of a mindfulness program with mindfulness-based interventions (MBI's) dedicated for adolescents with chronic pain.
  Interventions: Other: Mindfulness-based interventions (MBI's)

INTERVENTIONS:
Other: Mindfulness-based interventions (MBI's) — Mindfulness Based Intervention with eight sessions (one session per week) of two hours dedicated to adolescents will be provided. The intervention will focus on skill building and will incorporate mindfulness meditation, exercises and activities specially adapted to teenagers with chronic pain. Topics will include mind body connection, the effect of stress on pain, living in the present moment, focused awareness, responding versus reacting to pain and/ or difficult situations, non judgement, gratitude, kindness and compassion towards self and others.

SUMMARY:
The main objective is to study the feasibility of a program for the management of chronic painful adolescents in meditation groups. This program is an adaptation of the MBI-A (Mindfulness-based intervention for adolescent) program developed in another socio-cultural context (i.e. in Canada). The secondary objectives will be to study the effect of a mindfulness meditation program for adolescents on pain, quality of life, acceptance of pain, functional disability, catastrophism, anxiety-depression, emotional repercussions and acceptance of mindfulness

DETAILED DESCRIPTION:
Paediatric chronic pain can lead to serious consequences in terms of daily functioning (school absenteeism and loss of social interactions) and global quality of life. Mindfulness-based interventions (MBI's) approaches which emphasize acceptance rather than control of pain have gained increasing attention in adults with chronic pain. The effectiveness of MBI's for chronic pain in paediatric population remains largely unknown. An MBI program for adolescent was conducted in Toronto's Hospital for Sick Children and happened to be feasible and well received for adolescents with chronic pain conditions. The aim of the present program is to study the feasibility in France of a mindfulness program dedicated for adolescents with chronic pain.

An eight-session, two hour Mindfulness Based Intervention dedicated to adolescents will be provided. The intervention will focus on skill building and will incorporate mindfulness meditation, exercises and activities specially adapted to teenagers with chronic pain. Topics will include mind body connection, the effect of stress on pain, living in the present moment, focused awareness, responding versus reacting to pain and/ or difficult situations, non judgement, gratitude, kindness and compassion towards self and others.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers from 12 to 17 years of age followed at the Children's Hospital of Toulouse, as part of the Multidisciplinary Consultation of Pain
* including French.
* With the consent of the teenager and the parents
* Affiliated person or beneficiary of a social security scheme.

Exclusion Criteria:

* intellectual deficit not allowing to participate in a meditation program
* participating in research involving body therapies

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility in France of a mindfulness program : percentage of adolescents who will attend at least 6 of the 8 sessions | End of the mindfulness program (8 weeks)
  The primary outcome will be the percentage of adolescents who will attend at least 6 of the 8 sessions.

SECONDARY OUTCOMES:
Attendance rate | 1st session of the program (T1 week)
  Percentage of adolescents present at each program session
Attendance rate | 2nd session of the program (T2 weeks)
  Percentage of adolescents present at each program session
Attendance rate | 3rd session of the program (T3 weeks)
  Percentage of adolescents present at each program session
Attendance rate | 4th session of the program (T4 weeks)
  Percentage of adolescents present at each program session
Attendance rate | 5th session of the program (T5 weeks)
  Percentage of adolescents present at each program session
Attendance rate | 6th session of the program (T6 weeks)
  Percentage of adolescents present at each program session
Attendance rate | 7th session of the program (T7 weeks)
  Percentage of adolescents present at each program session
Attendance rate | 8th session of the program (T8 weeks)
  Percentage of adolescents present at each program session
Punctuality at the session | 1st session of the program (T1 week)
  binary criterion yes/no
Punctuality at the session | 2nd session of the program (T2 weeks)
  binary criterion yes/no
Punctuality at the session | 3rd session of the program (T3 weeks)
  binary criterion yes/no
Punctuality at the session | 4th session of the program (T4 weeks)
  binary criterion yes/no
Punctuality at the session | 5th session of the program (T5 weeks)
  binary criterion yes/no
Punctuality at the session | 6th session of the program (T6 weeks)
  binary criterion yes/no
Punctuality at the session | 7th session of the program (T7 weeks)
  binary criterion yes/no
Punctuality at the session | 8th session of the program (T8 weeks)
  binary criterion yes/no
Treatment acceptability | inclusion visit
  Rate of eligible adolescents who agreed to participate in the study
Treatment acceptability | 2nd session of the program (T2 weeks)
  Daily practice at home (binary criterion yes/no)
Treatment acceptability | 3rd session of the program (T3 weeks)
  Daily practice at home (binary criterion yes/no)
Treatment acceptability | 4th session of the program (T4 weeks)
  Daily practice at home (binary criterion yes/no)
Treatment acceptability | 5th session of the program (T5 weeks)
  Daily practice at home (binary criterion yes/no)
Treatment acceptability | 6th session of the program (T6 weeks)
  Daily practice at home (binary criterion yes/no)
Treatment acceptability | 7th session of the program (T7 weeks)
  Daily practice at home (binary criterion yes/no)
Treatment acceptability | 8th session of the program (T8 weeks)
  Daily practice at home (binary criterion yes/no)
Pain Level | Inclusion visit (baseline)
  Pain level will be assessed using Visual Analog Scale (from 0 "no pain" to 10 "the worst pain possible "). The pain will be measured by the average of the visual analogue rating scales evaluated over the last 8 days.
Pain Level | T2 Visit (1 week after the end of the 8-week program)
  Pain level will be assessed using Visual Analog Scale (from 0 "no pain" to 10 "the worst pain possible "). The pain will be measured by the average of the visual analogue rating scales evaluated over the last 8 days.
Pain Level | T3 Visit (3 months after the end of the 8-week program)
  Pain level will be assessed using Visual Analog Scale (from 0 "no pain" to 10 "the worst pain possible "). The pain will be measured by the average of the visual analogue rating scales evaluated over the last 8 days.
Quality of life at baseline : impact of adolescents health on their everyday life. | Inclusion visit (baseline)
  Quality of life will be assessed using the french scale VSPA-12 ("Vécu et Santé Perçue de l'adolescent (VSPA) - 12 items", "Lived and Health Perceived in 12 items) which is a self-questionnaire to assess the impact of adolescents health on their everyday life. The 12 items have five possible answers: never, rarely, sometimes, often, always.
Quality of life at the end of program | T2 Visit (1 week after the end of the 8-week program)
  Quality of life will be assessed using the french scale VSPA-12 ("Vécu et Santé Perçue de l'adolescent - 12 items", "Lived and Health Perceived in 12 items) which is a self-questionnaire to assess the impact of adolescents health on their everyday life. The 12 items have five possible answers: never, rarely, sometimes, often, always.
Quality of life in long term | T3 Visit (3 months after the end of the 8-week program)
  Quality of life will be assessed using the french scale VSPA-12 ("Vécu et Santé Perçue de l'adolescent - 12 items", "Lived and Health Perceived in 12 items) which is a self-questionnaire to assess the impact of adolescents health on their everyday life. The 12 items have five possible answers: never, rarely, sometimes, often, always.
Chronic pain acceptance | Inclusion visit (baseline)
  Chronic pain acceptance will be assessed using Chronic Pain Acceptance Questionnaire, Adolescent version (CPAQ-A) translated in French. CPAQ-A has 20 items For each item, the answer modalities are: 0= Never True, 1 = Rarely true, 2 = sometimes true, 3 = Often true, 4 = always true.
Chronic pain acceptance | T2 Visit (1 week after the end of the 8-week program)
  Chronic pain acceptance will be assessed using CPAQ-A (Chronic Pain Acceptance Questionnaire, Adolescent version) translated in French. CPAQ-A (Questionnaire for acceptance of chronic pain for adolescents) has 20 items For each item, the answer modalities are: 0= Never True, 1 = Rarely true, 2 = sometimes true, 3 = Often true, 4 = always true.
Chronic pain acceptance | T3 Visit (3 months after the end of the 8-week program)
  Chronic pain acceptance will be assessed using CPAQ-A (Chronic Pain Acceptance Questionnaire, Adolescent version) translated in French. CPAQ-A (Questionnaire for acceptance of chronic pain for adolescents) has 20 items For each item, the answer modalities are: 0= Never True, 1 = Rarely true, 2 = sometimes true, 3 = Often true, 4 = always true.
Functional disability | Inclusion visit (baseline)
  Functional disability will be assessed using FDI (Functional Disability Inventory) which is a functional disability scale to assess physical problems or any difficulties that adolescents may have in performing activities of daily living. FDI have 15 items. For each item, the answer modalities are 0 = no trouble, 1 = a little trouble, 2 = some trouble, 3 = a lot of trouble and 4 = impossible. The total FDI score is a sum of all of the items. The FDI score ranges from 0 to 60, with higher score indicating greater functional disability.
Functional disability | T2 Visit (1 week after the end of the 8-week program)
  Functional disability will be assessed using FDI (Functional Disability Inventory) which is a functional disability scale to assess physical problems or any difficulties that adolescents may have in performing activities of daily living. FDI have 15 items. For each item, the answer modalities are 0 = no trouble, 1 = a little trouble, 2 = some trouble, 3 = a lot of trouble and 4 = impossible. The total FDI score is a sum of all of the items. The FDI score ranges from 0 to 60, with higher score indicating greater functional disability.
Functional disability | T3 Visit (3 months after the end of the 8-week program)
  Functional disability will be assessed using FDI (Functional Disability Inventory) which is a functional disability scale to assess physical problems or any difficulties that adolescents may have in performing activities of daily living. FDI have 15 items. For each item, the answer modalities are 0 = no trouble, 1 = a little trouble, 2 = some trouble, 3 = a lot of trouble and 4 = impossible. The total FDI score is a sum of all of the items. The FDI score ranges from 0 to 60, with higher score indicating greater functional disability.
Anxiety and Depression | Inclusion visit (baseline)
  The anxiety and depression will be assessed using the french version of the Revised Children's Anxiety and Depression Scale (RCADS) intended to evaluate the symptomatology associated with anxiety disorders and major depression in children. This scale have 29 items. For each item, the possible answers are: never, sometimes, often, always.
Anxiety and Depression | T2 Visit (1 week after the end of the 8-week program)
  The anxiety and depression will be assessed using the french version of the Revised Children's Anxiety and Depression Scale (RCADS) intended to evaluate the symptomatology associated with anxiety disorders and major depression in children. This scale have 29 items. For each item, the possible answers are: never, sometimes, often, always.
Anxiety and Depression | T3 Visit (3 months after the end of the 8-week program)
  The anxiety and depression will be assessed using the french version of the Revised Children's Anxiety and Depression Scale (RCADS) intended to evaluate the symptomatology associated with anxiety disorders and major depression in children. This scale have 29 items. For each item, the possible answers are: never, sometimes, often, always.
Catastrophism | Inclusion visit (baseline)
  Catastrophism will be assessed using PCS-Ado (Pain Catastrophizing Scale for Francophone Adolescents) which identifies the thoughts and emotions that may be associated with the pain. PCS-Ado have 13 items. For each item, the possible answers are: never, rarely, sometimes, often and always.
Catastrophism | T2 Visit (1 week after the end of the 8-week program)
  Catastrophism will be assessed using PCS-Ado (Pain Catastrophizing Scale for Francophone Adolescents) which identifies the thoughts and emotions that may be associated with the pain. PCS-Ado have 13 items. For each item, the possible answers are: never, rarely, sometimes, often and always.
Catastrophism | T3 Visit (3 months after the end of the 8-week program)
  Catastrophism will be assessed using PCS-Ado (Pain Catastrophizing Scale for Francophone Adolescents) which identifies the thoughts and emotions that may be associated with the pain. PCS-Ado have 13 items. For each item, the possible answers are: never, rarely, sometimes, often and always.
Mindfulness acceptance | Inclusion visit (baseline)
  Mindfulness acceptance will be assessed using the French version of Five Facets Mindfulness Questionnaire (FFMQ) with 39 items. For each item the possible answers are: 1 = never or very rarely true, 2 = rarely true, 3 = sometimes true, 4 = often true, 5 = very often or always true.
Mindfulness acceptance | T2 Visit (1 week after the end of the 8-week program)
  Mindfulness acceptance will be assessed using the French version of Five Facets Mindfulness Questionnaire (FFMQ) with 39 items. For each item the possible answers are: 1 = never or very rarely true, 2 = rarely true, 3 = sometimes true, 4 = often true, 5 = very often or always true.
Mindfulness acceptance | T3 Visit (3 months after the end of the 8-week program)
  Mindfulness acceptance will be assessed using the French version of Five Facets Mindfulness Questionnaire (FFMQ) with 39 items. For each item the possible answers are: 1 = never or very rarely true, 2 = rarely true, 3 = sometimes true, 4 = often true, 5 = very often or always true.
Strengths and Difficulties | Inclusion visit (baseline)
  Strengths and difficulties will be assessed using the french version of the Strengths and Difficulties Questionnaire (SDQ-Fra) with 25 items. For each item, the possible answers are : not true, a little true, very true. The total difficulty score of the SDQ ranges from 0-40.
Strengths and Difficulties | T2 Visit (1 week after the end of the 8-week program)
  Strengths and difficulties will be assessed using the french version of the Strengths and Difficulties Questionnaire (SDQ-Fra) with 25 items. For each item, the possible answers are : not true, a little true, very true. The total difficulty score of the SDQ ranges from 0-40.
Strengths and Difficulties | T3 Visit (3 months after the end of the 8-week program)
  Strengths and difficulties will be assessed using the french version of the Strengths and Difficulties Questionnaire (SDQ-Fra) with 25 items. For each item, the possible answers are : not true, a little true, very true. The total difficulty score of the SDQ ranges from 0-40.
Adolescents satisfaction | T2 Visit (1 week after the end of the 8-week program)
  Adolescents satisfaction about the mindfulness program will be assessed using a satisfaction questionnaire with 8 items designed for this study. For each item, the modality answers are scored from 1 to 4.
Parents satisfaction | T2 Visit (1 week after the end of the 8-week program)
  Parents satisfaction about the mindfulness program followed by their children will be assessed using a satisfaction questionnaire with 8 items designed for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Agnès SUC, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hôpital des Enfants, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gray AR, Roberts CJ. The stability of resistance to diminazene aceturate and quihapyramine sulphate in a strain of Trypanosoma vivax during cyclical transmission through antelope. Parasitology. 1971 Aug;63(1):163-8. doi: 10.1017/s0031182000067512. No abstract available. PMID 5130089
- [Background] Simecek O, Kralik J. [Ethical justification of hemicorporectomy]. Rozhl Chir. 1973 Apr;52(4):240-3. No abstract available. Czech. PMID 4700163
- [Background] Bawa FL, Mercer SW, Atherton RJ, Clague F, Keen A, Scott NW, Bond CM. Does mindfulness improve outcomes in patients with chronic pain? Systematic review and meta-analysis. Br J Gen Pract. 2015 Jun;65(635):e387-400. doi: 10.3399/bjgp15X685297. PMID 26009534
- [Background] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Background] Zenner C, Herrnleben-Kurz S, Walach H. Mindfulness-based interventions in schools-a systematic review and meta-analysis. Front Psychol. 2014 Jun 30;5:603. doi: 10.3389/fpsyg.2014.00603. eCollection 2014. PMID 25071620
- [Background] Ruskin D, Harris L, Stinson J, Kohut SA, Walker K, McCarthy E. "I Learned to Let Go of My Pain". The Effects of Mindfulness Meditation on Adolescents with Chronic Pain: An Analysis of Participants' Treatment Experience. Children (Basel). 2017 Dec 15;4(12):110. doi: 10.3390/children4120110. PMID 29244734
- [Background] Ruskin DA, Gagnon MM, Kohut SA, Stinson JN, Walker KS. A Mindfulness Program Adapted for Adolescents With Chronic Pain: Feasibility, Acceptability, and Initial Outcomes. Clin J Pain. 2017 Nov;33(11):1019-1029. doi: 10.1097/AJP.0000000000000490. PMID 28328699
- [Result] Suc A, Cayzac D, Iannuzzi S, Garnier C, Bonneau B, Sommet A. Peacefull: A French mindfulness-based intervention for adolescents with chronic pain a feasibility study. Arch Pediatr. 2022 Nov;29(8):581-587. doi: 10.1016/j.arcped.2022.06.006. Epub 2022 Sep 13. PMID 36109288